CLINICAL TRIAL: NCT00103246
Title: Phase I Clinical Trial Using Topical Silicon Phthalocyanine (Pc 4) Photodynamic Therapy (PDT) for the Treatment of Pre-Malignant and Malignant Skin Conditions
Brief Title: Photodynamic Therapy Using Silicon Phthalocyanine 4 in Treating Patients With Actinic Keratosis, Bowen's Disease, Skin Cancer, or Stage I or Stage II Mycosis Fungoides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1Y04; P30CA043703 (NIH); CASE-CWRU-1Y04; 10-03-01 (Other: University Hospitals IRB); CASE1Y04 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2011-01

CONDITIONS: Lymphoma; Non-melanomatous Skin Cancer; Precancerous Condition
Keywords: skin cancer; squamous cell carcinoma of the skin; basal cell carcinoma of the skin; recurrent skin cancer; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; actinic keratosis; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Precancerous Conditions; Skin Neoplasms; Carcinoma, Basal Cell; Mycosis Fungoides; Sezary Syndrome; Keratosis, Actinic; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical silicon phthalocyanine 4 (Pc 4) + photodynamic therapy (Experimental): Topical silicon phthalocyanine 4 (Pc 4) followed by photodynamic therapy.
  Interventions: Drug: silicon phthalocyanine 4

INTERVENTIONS:
Drug: silicon phthalocyanine 4 — Participants receive topical silicon phthalocyanine 4 (Pc 4). One hour later, participants undergo photodynamic therapy. Treatment repeats weekly for up to 3 weeks (up to 3 total treatments for the same lesion OR up to 3 lesions treated if multiple lesions are present).Cohorts of 3 participants receive escalating doses of Pc 4 and visible light until the maximum tolerated dose (MTD) is determined.
  Other Names: Pc 4

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. Photodynamic therapy using silicon phthalocyanine 4 may be effective against skin cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of photodynamic therapy using silicon phthalocyanine 4 in treating participants with actinic keratosis, Bowen's disease, skin cancer, or stage I or stage II mycosis fungoides.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of photodynamic therapy using topically delivered silicon phthalocyanine 4 in participants with actinic keratosis, Bowen's disease, squamous cell or basal cell skin cancer, or stage IA, IB, IIA, or IIB mycosis fungoides.
* Determine the safety and toxicity of this therapy with emphasis on whether it induces photosensitivity in non-treated sites in these participants .
* Determine the antitumor mechanism of this therapy, by monitoring tissue changes via clinical, histological, immunohistochemical, and other biochemical markers, in these participants.
* Determine, preliminarily, the dose of this therapy that results in highest clearing rates in these participants.

OUTLINE: This is a dose-escalation study.

Participants receive topical silicon phthalocyanine 4 (Pc 4). One hour later, participants undergo photodynamic therapy. Treatment repeats weekly for up to 3 weeks (up to 3 total treatments for the same lesion OR up to 3 lesions treated if multiple lesions are present).

Cohorts of 3 participants receive escalating doses of Pc 4 and visible light until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 3 participants experiences dose-limiting toxicity. Three additional participants are treated at the MTD.

After completion of study therapy, participants are followed for up to 2 weeks.

PROJECTED ACCRUAL: A total of 16-45 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Actinic keratosis
  * Bowen's disease
  * Squamous cell skin cancer
  * Basal cell skin cancer
  * Clinical stage IA, IB, IIA, or IIB mycosis fungoides
* Fitzpatrick skin type I-IV

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patient must use effective contraception
* No diabetes mellitus
* No known hypersensitivity to ethanol or propylene glycol
* No significant history of photosensitivity, including diagnosis of any of the following:

  * Porphyria
  * Lupus erythematosus
  * Xeroderma pigmentosum
  * Severe polymorphous light eruption
  * Solar urticaria

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 2 weeks since prior anticancer radiotherapy
* No concurrent radiotherapy

Surgery

* Lesions must be healed after prior biopsy

Other

* More than 2 weeks since prior topical, local, or systemic anticancer therapy
* More than 2 weeks since prior anticancer phototherapy
* More than 2 weeks since prior photosensitizing medications, including any of the following:

  * Tetracyclines
  * Quinolones
  * Psoralens
  * Hydrochlorothiazide
  * Furosemide
  * Trimethoprim-sulfamethoxazole
  * Griseofulvin
  * Nalidixic acid
  * Amiodarone
  * Phenothiazines
  * High-dose nonsteroidal anti-inflammatory drugs
* No other concurrent photosensitizing medications
* No concurrent therapeutic dose of warfarin that may cause excessive bleeding during skin biopsy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Treatment repeats weekly for up to 3 weeks. Cohorts of 3 participants receive escalating doses of Pc 4 and visible light until the maximum tolerated dose (MTD) is determined.
Local toxicity as measured by physical exam and punch biopsy | at 24 hours and 2 weeks after the start of study treatment
Treatment efficacy as measured by physical exam and punch biopsy | at 24 hours and 2 weeks after the start of study treatment
Systemic photosensitivity as measured by minimum erythema dose (MED) testing | at 2, 24, and 48 hours after completion of photodynamic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Elma Baron, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States